CLINICAL TRIAL: NCT03144115
Title: Does Oxytocin Modulate Rewarding Effect of Metaphorical Compliments Fluctuating With Women's Fertility and Luteal Phase in a Romantic Context
Brief Title: Does Oxytocin Modulate Rewarding Effects in Women and Fluctuating Across the Menstrual Cycle
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-22
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: oxytocin; sex hormone; verbal reward; mate selection; metaphorical language
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- oxytocin fertility (Experimental): intranasal oxytocin administration (24IU) in women's fertility phase (LH>40 mIU/ml)
  Interventions: Drug: Oxytocin
- placebos fertility (Placebo Comparator): intranasal placebo administration (24IU) in women's fertility phase (LH>40 mIU/ml)
  Interventions: Drug: Placebos
- oxytocin luteal (Experimental): intranasal oxytocin administration (24IU) in women's luteal phase (LH<30 mIU/ml)
  Interventions: Drug: Oxytocin
- placebos luteal (Placebo Comparator): intranasal placebos administration (24IU) in women's luteal phase (LH<30 mIU/ml)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Oxytocin
  Other Names: oxytocin treatment
  Arms: oxytocin fertility; oxytocin luteal
Drug: Placebos
  Other Names: placebo control
  Arms: placebos fertility; placebos luteal

SUMMARY:
The aim of the study is to explore how the rewarding effect of men's verbal compliment is modulated by oxytocin and gonadal hormone in a romantic context.

DETAILED DESCRIPTION:
To investigate whether oxytocin (24IU) might interact with female sex hormone in modulating the rewarding effect of compliment to women in a romantic context.

The study employs a double-blind, within-subject, placebo-control design. Women will be administered with the same drug twice (oxytocin or placebo) respectively the fertile and luteal phase followed by a MRI scanning. During fMRI participants will rate men's attraction based on their facial pictures of average attractiveness associated with compliments of different combination of form and topic. Each male face will be paired with two sentences of the same kind. After the fMRI participants will recall the judgment followed by a memory test during which they have to indicate whether the they have seen the face during scanning (old) or whether it is an unknown face (new).

ELIGIBILITY:
Inclusion Criteria:

* Single in the past 3 months
* Healthy subjects with regular menstrual cycle

Exclusion Criteria:

* Pregnant, menstruating, taking oral contraceptives
* metal implanted, with tatoo, or hair dyed within 6 months
* participated in another intranasal experiment within 6 months
* with a history of past or current psychiatric or neurological disorder

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Oxytocin effect on neural activity as assessed via fMRI towards reward between fertility and luteal phases | 45min-120min after treatment
  Effects of oxytocin versus placebo nasal spray on neural processing of reward will be compared between different cycle phases

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of Chia, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Gao Z, Ma X, Zhou X, Xin F, Gao S, Kou J, Becker B, Kendrick KM. Oxytocin Reduces the Attractiveness of Silver-Tongued Men for Women During Mid-Cycle. Front Neurosci. 2022 Apr 28;16:760695. doi: 10.3389/fnins.2022.760695. eCollection 2022. PMID 35573309